CLINICAL TRIAL: NCT04618952
Title: The Effect of Calcium-D Supplements on the Blood Pressure of Postmenopausal Women, Myth or Reality ? A Triple-blind Randomized Clinical Trial
Brief Title: Effect of Calcium- D Supplement on Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1398.215
Record Dates: First submitted 2020-10-30; First posted 2020-11-06 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Hypertension
Keywords: hypertension; calcium-D; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group A and group B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment (Active Comparator): patients received calcium D
  Interventions: Drug: Calcium D
- control (Placebo Comparator): patients received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium D — calcium D supplementation given to postmenopausal females
  Arms: treatment
Drug: Placebo — Placebo
  Arms: control

SUMMARY:
Triple-blind randomized clinical trial was done on 98 hypertensive women of postmenopausal ages in 2019. The study was executed for 8 weeks with close follow up and , 24-hour Ambulatory blood pressure monitoring (ABPM) was used to record the initial and final blood pressures of all participants. Patients were randomized to calcium-D supplement and placebo

DETAILED DESCRIPTION:
Triple-blind randomized clinical trial were performed on 98 hypertensive women of postmenopausal ages in 2019. They were randomly divided into a control group of 50 members and a treatment group of 48 members. Randomization was based on block randomization method with block size=2 and ratio 2:2 for drug and placebo. To achieve triple blinding, patients were divided into "A" and "B" groups(by the mentioned randomization method). "A" was assigned to treatment and "B" to placebo but this assignment was not revealed to the patients, trial conductors and result assessors till the end of data analysis.

Oral calcium-D supplements were given to the treatment group in the form of tablets named Vana Flex® from Vana Darou Gostar Co. (VDG Co.). Each tablet contained 500 milligrams of calcium carbonate and 200 international units (IU) of vitamin D3(cholecalciferol). The placebo pills for the control group were chose in a way that looked similar to the calcium-D tablets in shape and color. The placebo tablets we used in this trial were made up of magnesium stearate 0.2 %, starch 10%, avicel 30%, and lactose 60%. The calcium-D and placebo tablets were both packed identically in order to assure blindness and the patients were told to take one tablet per day. The treatment and placebo group started drugs beside their previous hypertension medications.

24-hour Ambulatory blood pressure monitoring (ABPM) was done primarily for all of the participants to record the initial blood pressure of patients and after completion of study period

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal female with hypertension
* receiving antihypertensive drugs

Exclusion Criteria:

* history of coronary artery disease
* congestive heart failure
* chronic renal disease
* hypercalcemia
* nephrolithiasis
* any other contraindications of calcium use

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal female
Enrollment: 98 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure in 24 hours | 60 days
  24 hour holter monitoring was used to measure systolic blood pressure in automated measurement for 80 times at home, in millimeter of mercury and device reported the mean of these systolic pressures
Mean diastolic blood pressure in 24 hours | 60 days
  24 hour holter monitoring was used to measure diastolic blood pressure in automated measurement for 80 times at home, in millimeter of mercury and device reported the mean of these diastolic pressures
Blood pressure dipping at night | 60 days
  24 hour holter monitoring was used to measure mean systolic blood pressure in automated measurement for 80 times at home, in millimeter of mercury and device reported the mean of these systolic pressures, and comparing mean of systolic blood pressure at night and day, and dippers are those who have more than 10% drop in mean systolic blood pressure at nigh

SECONDARY OUTCOMES:
Effect of amlodipine on the effect of calcium-D supplements | 60 days
  patients in study divided to two groups ,who received amlodipine or not and effect of calcium-D supplement, was compared between these two groups, by 24 hour holter monitoring of blood pressure

CONTACTS AND LOCATIONS:
Locations (3):
- Iran (3):
  - Professor Kojuri cardiology clinic, Shiraz, Fars
  - Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars
  - Education Developmen Center, Shiraz, Fars

IPD SHARING:
Plan to Share IPD: No
Results and article will be available

REFERENCES:
- [Derived] Sharifi F, Heydarzadeh R, Vafa RG, Rahmani M, Parizi MM, Ahmadi A, Zamiri B, Montaseri M, Kojuri J. The effect of calcium and vitamin D supplements on blood pressure in postmenopausal women: myth or reality? Hypertens Res. 2022 Jul;45(7):1203-1209. doi: 10.1038/s41440-022-00930-3. Epub 2022 May 13. PMID 35562420